CLINICAL TRIAL: NCT02678728
Title: Effect of Intraoperative Dexmedetomidine on Lung Protection Following Thoracic Aorta Surgery With Hypothermic Circulatory Arrest: a Randomized Clinical Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Young Song, Associate Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 3-2015-0252
Record Dates: First submitted 2016-01-19; First posted 2016-02-10 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Chronic Dissecting Aneurysm of Thoracic Aorta; Chronic Nontraumatic Dissection of Thoracic Aorta; Dissecting Aneurysm of the Thoracic Aorta
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Experimental): 1ug/kg IV loading over 20 minutes followed by 0.5ug/kg/hr IV infusion until 12hr of aortic cross clamp off
  Interventions: Drug: Dexmedetomidine
- Normal saline (Placebo Comparator): IV loading and infusion of same volume of normal saline after induction until 12hr of aortic cross clamp off
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — 1ug/kg IV loading over 20 minutes followed by 0.5ug/kg/hr IV infusion until 12 hrs of aortic cross clamp off
  Other Names: precedex
  Arms: Dexmedetomidine
Drug: normal saline — IV loading and infusion of same volume of normal saline after induction until 12 hrs of aortic cross clamp off
  Arms: Normal saline

SUMMARY:
Dexmedetomidine has been known to protect the lung against inflammation and oxidative stress in diverse clinical settings. The investigators aimed to investigate the lung protective effect of dexmedetomidine in patients undergoing thoracic aortic surgery with hypothermic circulatory arrest, which is associated with systemic inflammatory response, and oxidative stress.

DETAILED DESCRIPTION:
Patients will be divided into 2 groups; dexmedetomidine group and control group. Dexmedetomidine group will receive dexmedetomidine during and after thoracic artery surgery. And control group will receive the same amount of normal saline instead. Analyzing patients lung function and serum factors, which indicates the degree of systemic inflammatory responses and oxidative stress, The investigators will investigate the protective effect of dexmedetomidine on lung.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing thoracic aorta surgery with hypothermic circulatory arrest, over 20-of age

Exclusion Criteria:

* Unstable vital sign before surgery
* Severe pulmonary disease requiring consistent treatment
* Illiterate
* Pregnancy

Ages: 20 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-02-28 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Changes of lung oxygenation from baseline to 24 hr after reperfusion | after induction of anesthesia / after reperfusion 1hr / after reperfusion 6hr / after reperfusion 12hr / after reperfusion 24hr
  Lung oxygenation will be assessed by arterial blood gas analysis
Changes of lung compliance from baseline to 24 hr after reperfusion | after induction of anesthesia / after reperfusion 1hr / after reperfusion 6hr / after reperfusion 12hr / after reperfusion 24hr
  Lung compliance will be displayed on the ventilator

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No